CLINICAL TRIAL: NCT01189630
Title: Medtronic Observational Study in the "Real World" of Implantable Electronic Cardiac Devices
Acronym: OBSERVE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medtronic Comercial Ltda. (Industry)
Responsible Party: Roberto Takeda, Medtronic Comercial
Other Study IDs: MDT-01-2010
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Heart Failure
Keywords: "Real World" Electronic Database with clinical information; related to Implantable Cardiac devices.
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Observational Study in the "Real World" of Implantable Electronic Cardiac Devices will enable the construction of an electronic database with local access to clinical information, which will collect and disseminate epidemiologic data on demography, cardiovascular mortality and morbidity, and potential risk factors for a selected group of patients. These clinical variables will be analyzed against the data, as based in the programming of devices and the diagnostics. Approved descriptive statistics and analyses will be made available via Internet. The study will describe statistical indexes on sub-groups representing more than 10% of total of datasets.

The study will be open to include any patient that had a Medtronic electronic device implanted, pacemakers, ICD, ICD with CRP. The study will be also adapted for devices implanted in the present and for devices to be implanted in patients in the future.

DETAILED DESCRIPTION:
This study is a Prospective, Multicenter Observational Post Market Release Study. It shall involve around 2,000 patients that are eligible for Implantable Cardiac Pacemakers (IPG) implantation, 500 patients eligible for Cardiac Resynchronization Pacemakers (CRT-P) implantation, 1,000 patients eligible for the implantation of Implantable Cardioverter Defibrillators with or without Cardiac Resynchronization Pacemakers (CDI, CRT-D), and around 20 centers in Brazil. Patients will be consecutively enrolled in centers among those selected for the implantation of a Medtronic device in accordance with indications approved.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than18 years of age
* Patient agrees to participate in the study and is able to sign the Data Release Form
* High probability of adherence to follow-up requirements

Exclusion Criteria:

* Patients who want to be enrolled in another clinical study during at the same time that he/she is part of OBSERVE study.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible to participate in this study are among those having an approved indication for the implantation of Implantable Cardiac Pacemakers (IPG), Cardiac Resynchronization Pacemakers (CRT-P), Implantable Cardioverter Defibrillator (ICD) with or without Cardiac Resynchronization Pacemakers (CRT-D).
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2010-12; Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Takeda, MD, Study Director — Medtronic Comercial
Locations (1):
- Medtronic Comercial, São Paulo, São Paulo, Brazil